CLINICAL TRIAL: NCT01032434
Title: An 8-week, Open-label Study to Evaluate the Effect of Sertraline on Polysomnogram in Depressive Patients With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang Dong Provincial Mental Health Institute (Other)
Responsible Party: Principal Investigator, Bin Zhang, Sleep Centre, Guang Dong Provincial Mental Health Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WS 458774
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Depression
Keywords: sertraline; Polysomnograph
MeSH Terms: conditions — Depression | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sertraline (Experimental): sertraline: 50-200mg/day
  Interventions: Drug: sertraline

INTERVENTIONS:
Drug: sertraline — sertraline: 50-200mg/day
  Other Names: zoloft

SUMMARY:
Major depressive disorder is associated with several sleep Polysomnograph (PSG) findings: (1) impaired sleep continuity; (2) non-REM (NREM) changes; and (3) enhanced rapid eye movement (REM) sleep. The first two patterns are common in other psychiatric disorders, while the REM pattern is very characteristic in depression, so the phase-advance theory was accepted by most of psychiatrists. Many researchers have focused on the biological rhythm to investigate the etiological and pathophysiology of depression, and they think depression can be cured if its sleep abnormality is ameliorated.

It is well known that most of antidepressants treat depression through 5-hydroxytryptamine (5-HT) neurons. 5-HT also affects the regulation of the sleep-wake cycle and the sleep microarchitecture. Many all-night PSG studies have shown tricyclic antidepressants can ameliorate the sleep architecture abnormality in depression by producing rapid suppression of REM sleep.

Compared to TCAs, SSRIs are generally less sedating because of its high selectivity for serotonin receptors. SSRIs can suppress REM sleep and delay REM latency too, but they increase awakenings and reduce SWS at the same time. One PSG study shown sertraline minimally increases sleep efficiency and reduces nocturnal wakefulness time, which may benefit depressive patients. However, this study compared the sleep architecture before and after 12 weeks of pharmacotherapy, so the tolerance to the disturbance of sleep architecture in antidepressants appears to develop over several weeks of treatment. Sertraline has a greater potency against 5-HT reuptake as well as better selectivity for 5-HT reuptake relative to NE reuptake than any other SSRIs, and the relative selectivity of sertraline for inhabiting 5-HT reuptake relative to DA reuptake is somewhat less than of any other SSRIs. So it has chance to exhibit better effect on sleep architecture in depressive patients.

Finally, it is difficult to be determined that the unique phenomenon of sertraline is its genuine characteristics or the tolerance after 12-week treatment, so it is crucial to assess the effect of sertraline on sleep architecture in acute treatment. We hypothesized that sertraline could suppress the REM sleep, and have little damage to the sleep architecture of depressive patient.

DETAILED DESCRIPTION:
[Abstract] Purpose of the study: To evaluate the effect of sertraline on polysomnographic (PSG) variables and clinical improvement in the treatment of depressive patients with insomnia. Methods used: The study design was 8-week and open-label trial. Patients were diagnosed as major depressive disorder. Their Hamilton Rating Scale for Depression (HRSD) score was more than 18, and HRSD-sleep disturbance score was more than 3. After 7-day wash-out period and 2 nights PSG (the first night as adaptive and the second night as baseline), 31 depressive patients were administered by sertraline as 50 mg in 8 am in the 1st day. The dosage of sertraline would be titrated during the 8-week treatment, and the maximum was lower than 200 mg/day. The primary endpoints were the changes of PSG variables from baseline to the 56th Day. The secondary endpoints were the changes of subjective sleep quality and clinical performance from baseline to the 56th Day. Their sleep quality was evaluated with Epworth Sleepiness Scale (ESS) and Pittsburgh Sleep Quality Index (PSQI), and their clinical performance was evaluated with HRSD and Clinical Globe Impression (CGI). Summary of results containing real data and appropriate statistical assessments: The Intent-to-Treat analysis included 31 subjects. The final dosage was titrated as 130.6±47.8 mg/day. The Rapid Eye Movement (REM) sleep latency was prolonged significantly in the 1st day and throughout 8-week treatment. The percentage of REM sleep decreased significantly in the 1st day, but increased gradually along the following treatment. AI reached the highest level in the 1st day (13.8±7.2), and decreased along the following treatment. SL decreased significantly and reached normal range (<30minutes) after the visit of 14th day. The percentage of stage 3 increased gradually, and became higher in the 14th, 28th, 56th days. HRSD score was similar between baseline and the 1st day, and became significantly lower in the 14th, 28th, and 56th day. Similar pattern was shown in CGI. Scores of HRSD-sleep disturbance, PSQI, ESS decreased gradually throughout the treatment. The sleep latency in multiple sleep latency test maintained stable throughout treatment. The reducing score rates of HRSD and CGI-GI significantly correlated with the reducing score rate of REM latency in all visits, and they also significantly correlated with sleep latency, sleep efficiency, and stage 3 in some visits. Further, significant correlation was shown between the reducing score rate of HRSD in the 56th day and the the reducing score rate of REM latency in the 1st day (r=-0.733, P=0.003). Conclusions: Sertraline was an effective antidepressant, and its effectiveness had relationship with the reduction of REM latency during the 8-week treatment. Further, the final clinical improvement could be predicted by the extent of shorten REM latency in the first night. So the suppression of REM sleep might be the key mechanism of antidepressive[1]. On the other hand, Sertraline had little alerting property without sleep disturbance in the treatment[2]. This property of sertraline must benefit the remission of depression, and the remission contributed the sleep improvement in turn. It was virtuous cycle in depressive treatment.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study patients must fulfil all of the following criteria:

1. Provision of written informed consent by patient or his/her legal guardian
2. Hospitalised for a diagnosis of major depressive disorder by DSM-IV (296.2X, 296.3X)
3. HRSD score>18
4. Total score of sleep disturbance factor in HRSD (items 4, 5, and 6; score range, 0-6)>3
5. Females or males, and aged 18 to 65 years
6. Able to understand and comply with the requirements of the study

Exclusion Criteria:

Any of the following is regarded as a criterion for exclusion from the study:

1. Pregnancy or lactation
2. Any DSM-IV Axis I disorder, except for major depressive disorder
3. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
4. Known intolerance or lack of response to sertraline, as judged by the investigator
5. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
6. Use of any of the following cytochrome P450 3A4 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
7. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
8. Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
9. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment
10. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
11. Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension) as judged by the investigator
12. Organic change was founded by brain CT
13. Involvement in the planning and conduct of the study
14. Previous enrolment or randomisation of treatment in the present study
15. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
16. An absolute neutrophil count (ANC) of 1.5 x 109/L
17. Sleep disorder such as Apnea and Hyponea Syndrome, PLMS and narcolepsy
18. The work time is rotate and/or often flies across the time zone
19. Concomitant use in patients taking monoamine oxidase inhibitors (MAOIs)
20. Concomitant use in patients taking pimozide

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
the effect of sertraline on suppressing the percentage of REM sleep in depressive patients with insomnia as mono-therapy | 56 days

SECONDARY OUTCOMES:
the effect of sertraline on sleep continuity and SWS as mono-therapy | 56 days
the correlation between the degree of REM suppression with the degree of clinical improvement in the treatment of sertraline as mono-therapy. | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Bin Zhang, M.D&Ph.D, Principal Investigator — Guang Dong Provincial Mental Health Institute
Locations (1):
- Guangdong Provincial Mental Health Institute, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhang B, Hao Y, Jia F, Tang Y, Li X, Liu W, Arnulf I. Sertraline and rapid eye movement sleep without atonia: an 8-week, open-label study of depressed patients. Prog Neuropsychopharmacol Biol Psychiatry. 2013 Dec 2;47:85-92. doi: 10.1016/j.pnpbp.2013.08.010. Epub 2013 Aug 29. PMID 23994660